CLINICAL TRIAL: NCT01662440
Title: A Phase III, Multicenter, Observer-blind, Safety and Immunogenicity Study of Rabies Vaccine and Japanese Encephalitis Vaccine Administered Concomitantly and/or Separately According to 1 of 2 Different Preexposure Prophylaxis Schedules to Healthy Adult Subjects.
Brief Title: Safety and Immunogenicity of 2 Different Vaccination Schedules of Rabies and Japanese Encephalitis Vaccines in Healthy Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V49_23; 2011-005173-23 (EudraCT Number)
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Rabies; Japanese Encephalitis
Keywords: Rabies; JE; accelerated schedule
MeSH Terms: conditions — Rabies; Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- R/JE - Conv (Active Comparator): Subjects received Rabies and Japanese Encephalitis (JE) vaccines following the conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
  Interventions: Biological: Rabies; Biological: Japanese Encephalitis; Other: Placebo
- R/JE - Acc (Experimental): Subjects received Rabies and JE vaccines following the accelerated schedule, ie, Rabies vaccination on days 1, 4, and 8, and placebo on day 29 in the right arm or leg; and JE vaccination on days 1 and 8, and placebo on day 29 in the left arm.
  Interventions: Biological: Rabies; Biological: Japanese Encephalitis; Other: Placebo
- R - Conv (Active Comparator): Subjects received Rabies vaccine following the conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and placebo on days 1, 8 and 29 in the left arm.
  Interventions: Biological: Rabies; Other: Placebo
- JE - Conv (Active Comparator): Subjects received JE vaccine following the conventional schedule, ie, placebo on days 1, 4, 8 and 29 in the right arm or leg; and JE vaccination on days 1 and 29 and placebo injection on day 8 in the left arm.
  Interventions: Biological: Japanese Encephalitis; Other: Placebo

INTERVENTIONS:
Biological: Rabies — Subjects received three doses of Rabies, whole virus vaccine (inactivated, Germany).
  Arms: R - Conv; R/JE - Acc; R/JE - Conv
Biological: Japanese Encephalitis — Subjects received two doses of Japanese Encephalitis vaccine.
  Arms: JE - Conv; R/JE - Acc; R/JE - Conv
Other: Placebo — Subjects received either two, three, four or five doses of normal saline, 0.9% w/v sodium chloride depending on the vaccine group.

SUMMARY:
Establish non-inferiority of the immune response and evaluate the safety and tolerability of Rabies and Japanese Encephalitis (JE) vaccines given concomitantly or alone and according to either of 2 schedules for preexposure prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 65 years of age (inclusive).
2. Subjects who have given written consent.
3. Individuals in good health as per investigator judgement.

Exclusion Criteria:

1. If female, pregnancy or unwillingness to practice acceptable contraception.
2. If female, pregnant or breast-feeding or any positive/indeterminate pregnancy test.
3. Contraindication or precaution against Rabies and Japanese Encephalitis vaccination.
4. Unable to comprehend and to follow all required study procedures for the whole period of the study.
5. Participating in any other clinical trial 30 days prior to first study visit.
6. History of previous rabies/rabies immunoglobulin and/or Japanese Encephalitis immunization.
7. Receiving or planning to receive anti-malarial medications (e.g. Mefloquine) 14 days prior to Day 1 vaccination through Day 43.
8. Received any other vaccines within 2 weeks prior to enrollment in this study or plan to receive any vaccine within 4 weeks from the study vaccines.
9. Ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.
10. Individuals who are part of study personnel or close family members conducting this study.
11. Body temperature ≥38 degrees Celsius (≥ 100.4° F) within 3 days of intended study vaccination.
12. Plans to travel within the next year to areas where Rabies and/or Japanese Encephalitis vaccine may be considered or offered. This includes but is not limited to India, Asia, Pacific-Rim, African countries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (3):
- Institute of Specific Prophylaxis and Tropical Medicine Center for Pathophysiology, Infectious Diseases and Immunology Medical University of Vienna, Kinderspitalgasse 15, Vienna, Austria
- Bernhard Nocht Institute for Tropical Medicine, Bernhard-Nocht-Strasse 74, Hamburg, Germany
- The University of Zurich, Rämistrasse 71, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Cramer JP, Jelinek T, Paulke-Korinek M, Reisinger EC, Dieckmann S, Alberer M, Buhler S, Bosse D, Meyer S, Fragapane E, Costantini M, Pellegrini M, Lattanzi M, Dovali C. One-year immunogenicity kinetics and safety of a purified chick embryo cell rabies vaccine and an inactivated Vero cell-derived Japanese encephalitis vaccine administered concomitantly according to a new, 1-week, accelerated primary series. J Travel Med. 2016 Mar 19;23(3):taw011. doi: 10.1093/jtm/taw011. Print 2016 Mar. PMID 26994987
- [Derived] Jelinek T, Cramer JP, Dieckmann S, Hatz C, Paulke-Korinek M, Alberer M, Reisinger EC, Costantini M, Gniel D, Bosse D, Lattanzi M. Evaluation of rabies immunogenicity and tolerability following a purified chick embryo cell rabies vaccine administered concomitantly with a Japanese encephalitis vaccine. Travel Med Infect Dis. 2015 May-Jun;13(3):241-50. doi: 10.1016/j.tmaid.2015.05.008. Epub 2015 May 18. PMID 26005163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from five sites in Germany, one site in Austria, and one site in Switzerland.
Pre-assignment Details: All subjects were included in the trial.
Groups:
- R/JE - Conv: Subjects received Rabies and Japanese Encephalitis (JE) vaccines, conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
- R/JE - Acc: Subjects received Rabies and JE vaccines, accelerated schedule, ie, Rabies vaccination on days 1, 4, and 8, and placebo on day 29 in the right arm or leg; and JE vaccination on days 1 and 8, and placebo on day 29 in the left arm.
- R - Conv: Subjects received Rabies vaccine, conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and placebo on days 1, 8 and 29 in the left arm.
- JE - Conv: Subjects received JE vaccine, conventional schedule, ie, placebo on days 1, 4, 8 and 29 in the right arm or leg; and JE vaccination on days 1 and 29 and placebo injection on day 8 in the left arm.
Period: Overall Study
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv
Started | 167 | 217 | 221 | 56
Completed | 158 | 211 | 215 | 52
Not Completed | 9 | 6 | 6 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 4 | 1
Not completed — Subject moved to another country. | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- R/JE - Conv: Subjects received Rabies and JE vaccines, conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
- Total: Total of all reporting groups
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv | Total
Number analyzed (Participants) | 167 | 217 | 221 | 56 | 661
Age, Continuous [Mean (Standard Deviation); unit: year] | 37.3 (13.4) | 36.8 (12.7) | 35.7 (12.6) | 38.8 (13.3) | 36.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 128 | 125 | 30 | 359
  Male | 91 | 89 | 96 | 26 | 302

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With RVNA Concentrations ≥0.5 IU/mL At 7 Days After Last Active Vaccination
Description: Immune response was measured as the percentage of subjects with rabies virus neutralizing antibody (RVNA) concentrations ≥0.5 IU/mL, evaluated using the rapid fluorescent focus inhibition test at day 7 after last active vaccination, i.e. the third out of four vaccinations given in the accelerated Rabies vaccine schedule and the fourth out of four vaccinations given in the conventional Rabies vaccine schedule.
  As per study design, this primary immunogenicity outcome measure aimed to demonstrate non-inferiority of R/JE - Acc Vs R - Conv.
Time Frame: Day 7 after last active vaccination (day 15 - group that received accelerated schedule, day 36 - group that received conventional schedule)
Population: Analysis was done on the per-protocol (PP) dataset, ie, the subjects who received the vaccine correctly, provided evaluable serum samples at the relevant time points, and had no major protocol violations as defined prior to unblinding.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- R/JE - Acc: Subjects received Rabies and JE vaccines, accelerated schedule, ie, Rabies vaccination on days 1, 4, and 8, and placebo on day 29 in the right arm or leg, and JE vaccination on days 1 and 8, and placebo on day 29 in the left arm.
- R - Conv: Subjects received Rabies vaccine, conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg, and placebo on days 1, 8 and 29 in the left arm.
Arm/Group | R/JE - Acc | R - Conv
Number analyzed (Participants) | 209 | 207
Percentages of subjects | 100 [97 to 100] | 100 [97 to 100]
Statistical Analysis 1: Comparison: R/JE - Acc vs R - Conv; To establish non-inferiority of the immune response of Rabies vaccine (administered concomitantly with JE vaccine) accelerated schedule as compared to conventional schedule at 7 days after last active vaccination; Test type: Non-Inferiority or Equivalence — The immune response of accelerated schedule of the Rabies vaccine considered non-inferior to the conventional schedule if the lower bound of the two-sided 97.5% Confidence Intervals (CI) of the difference in the percentages of subjects with RVNA titer ≥0.5 IU/mL measured 7 days after last active vaccination is greater than -5; Difference in percentages of subjects = 0, 97.5% CI 2-sided [-2.8 to 2.8]

2. Primary Outcome: Percentages of Subjects With PRNT50 Titer ≥1:10 At 28 Days After Last Active Vaccination
Description: Immune response was measured as the percentages of subjects with a titer of ≥1:10 in a 50% plaque reduction neutralization test (PRNT50) 28 days after last active vaccination, ie, the second out of three vaccinations given in the accelerated JE vaccine schedule and the third out of three vaccinations given in the conventional JE vaccine schedule.
  As per study design, this primary immunogenicity outcome measure aimed to demonstrate non-inferiority of R/JE - Acc Vs JE - Conv.
Time Frame: Day 28 after last active vaccination (day 36 - group that received accelerated schedule, day 57 - group that received conventional schedule)
Population: Analysis was done on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- JE - Conv: Subjects received JE vaccine, conventional schedule, ie, placebo on days 1, 4, 8 and 29 in the right arm or leg, and JE vaccination on days 1 and 29 and placebo injection on day 8 in the left arm.
Arm/Group | R/JE - Acc | JE - Conv
Number analyzed (Participants) | 209 | 49
Percentages of subjects | 99 [96 to 100] | 100 [93 to 100]
Statistical Analysis 1: Comparison: R/JE - Acc vs JE - Conv; Non-inferiority of the immune response of JE vaccine (administered concomitantly with Rabies vaccine) accelerated schedule as compared to conventional schedule at 28 day after last active vaccination; Test type: Non-Inferiority or Equivalence — The immune response of accelerated schedule of the JE vaccine is considered non-inferior to the conventional schedule if the lower bound of the two-sided 97.5% CI of the difference in the percentages of subjects with PRNT50 titer ≥1:10 measured 28 days after last active vaccination is greater than -10; Difference in percentages of subjects = -1, 97.5% CI 2-sided [-4.8 to 7.9]

3. Secondary Outcome: RVNA Geometric Mean Concentrations (GMCs) At 28 Days After Last Active Vaccination
Description: Immune response was measured as the RVNA GMCs 28 days after last active vaccination, ie, day 57 for all groups that received the conventional schedule.
  Data were adjusted using ANOVA model, as per protocol specification.
Time Frame: Day 57 (28 days after last active vaccination)
Population: Analysis was done on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- R/JE - Conv: Subjects received Rabies and JE vaccines, conventional schedule, ie, Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg, and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
Arm/Group | R/JE - Conv | R - Conv
Number analyzed (Participants) | 157 | 204
IU/mL | 11 [9 to 12] | 9.9 [8.57 to 11]
Statistical Analysis 1: Comparison: R/JE - Conv vs R - Conv; Non-inferiority of the immune response of Rabies vaccine (administered concomitantly with JE vaccine) as compared to Rabies vaccines (administered alone) as given according to conventional schedule at 28day after last active vaccination; Test type: Non-Inferiority or Equivalence — The conventional schedule of Rabies vaccine co-administered with JE vaccine considered non inferior to the conventional schedule of Rabies vaccine administered alone if the lower bound of the two-sided 95% CI of the ratio of GMCs measured 28 days after last active vaccination is greater than 0.667; Between groups ratio of GMCs = 1.07, 95% CI 2-sided [0.86 to 1.32]

4. Secondary Outcome: PRNT50 Geometric Mean Titers (GMTs) At 28 Days After Last Active Vaccination
Description: Immune response was measured as the PRNT50 GMTs 28 days after last active vaccination, ie, day 57 for all groups that received the conventional schedule.
  Data were adjusted using ANOVA model, as per protocol specifications.
Time Frame: Day 57 (28 days after last active vaccination)
Population: Analysis was done on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- JE - Conv: Subjects received JE vaccine, conventional schedule, i.e. placebo on days 1, 4, 8 and 29 in the right arm or leg; and JE vaccination on days 1 and 29 and placebo injection on day 8 in the left arm.
Arm/Group | R/JE - Conv | JE - Conv
Number analyzed (Participants) | 157 | 49
Titers | 291 [256 to 331] | 331 [265 to 415]
Statistical Analysis 1: Comparison: R/JE - Conv vs JE - Conv; Non-inferiority of the immune response of JE vaccine (administered concomitantly with Rabies vaccine) as compared to JE vaccine (administered alone) as given according to conventional schedule at day 28 after last active vaccination; Test type: Non-Inferiority or Equivalence — The conventional schedule of JE vaccine co-administered with Rabies vaccine considered non inferior to the conventional schedule of JE vaccine administered alone if the lower bound of the two-sided 95% CI of the ratio of GMTs measured 28 days after last active vaccination is greater than 0.5; Ratio of GMTs = 0.88, 95% CI 2-sided [0.68 to 1.13]

5. Secondary Outcome: Percentages of Subjects With RVNA Concentrations ≥0.5 IU/mL At 28 Days After Last Active Vaccination
Description: Immune response was measured as the percentages of subjects with RVNA concentration ≥0.5 IU/mL 28 days after last active vaccination, ie, day 36 for the group that received the accelerated schedule and day 57 for the group that received the conventional schedule.
  As per study design, this secondary immunogenicity outcome measure aimed to demonstrate non-inferiority of R/JE - Acc Vs R - Conv.
Time Frame: Day 36 and day 57 (28 days after last active vaccination)
Population: Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | R/JE - Acc | R - Conv
Number analyzed (Participants) | 206 | 204
Percentages of subjects | 99 [96 to 100] | 100 [97 to 100]
Statistical Analysis 1: Comparison: R/JE - Acc vs R - Conv; Non-inferiority of the Rabies immune response (administered concomitantly with JE vaccine) as given according to an accelerated schedule as compared Rabies vaccine (administered alone) as given to a conventional schedule at day 28 after last active vaccination; Test type: Non-Inferiority or Equivalence — The immune response of accelerated schedule of the Rabies vaccine is considered non-inferior to the Rabies vaccine conventional schedule if the lower bound of the two-sided 95% CI of the difference in the percentages of subjects with RVNA titer ≥0.5 IU/mL measured 28 days after last active vaccine administration is greater than -5; Difference in percentages of subjects = -1, 95% CI 2-sided [-3.8 to 1.4]

6. Secondary Outcome: Percentage of Subjects With PRNT50 Titer ≥1:10 At 7 Days After Last Active Vaccination
Description: Immune response was measured as the percentage of subjects with PRNT50 titer of ≥1:10 7 days after last active vaccination, ie, day 15 for the group that received the accelerated schedule and day 36 for the group that received the conventional schedule.
  As per study design, this secondary immunogenicity outcome measure aimed to demonstrate non-inferiority of R/JE - Acc Vs JE - Conv.
Time Frame: Day 15 and day 36 (28 after last active vaccination)
Population: Analysis was done on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- JE - Conv: Group Description Subjects received Rabies and JE vaccines, conventional schedule, i.e. Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
Arm/Group | R/JE - Acc | JE - Conv
Number analyzed (Participants) | 209 | 47
Percentages of subjects | 99 [96 to 100] | 100 [92 to 100]
Statistical Analysis 1: Comparison: R/JE - Acc vs JE - Conv; Non-inferiority of the immune response of JE vaccine (administered concomitantly with Rabies vaccine) as given according to an accelerated schedule as compared to JE vaccine (administered alone) as given according to a conventional schedule at 7day after last active vaccine administration; Test type: Non-Inferiority or Equivalence — The immune response of accelerated schedule of the JE vaccine considered non-inferior to the conventional schedule if the lower bound of the two-sided 95% CI of the difference in the percentages of subjects with PRNT50 titer ≥1:10 measured 7 days after last active vaccine administration is greater than -10; Difference in percentages of subjects = -1, 95% CI 2-sided [-4.1 to 6.2]

7. Secondary Outcome: Kinetics of Rabies Immune Response Measured as Percentage of Subjects With RVNA Concentration ≥0.5 IU/mL
Description: To evaluate the kinetics of antibody response to Rabies vaccine, the immunogenicity was measured as the percentage of subjects with RVNA concentrations ≥0.5 IU/mL on days 1, 8, 15, 36, 57, 91, 181, and 366.
Time Frame: Day 1, 8, 15, 36, 57, 91, 181 and Day 366
Population: Analysis was done on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv
Number analyzed (Participants) | 166 | 215 | 218
Percentages of subjects
  Day 1 | 1 [0.015 to 3] | 1 [0 to 3] | 1 [0 to 4]
  Day 8 (N=161, 210, 213) | 4 [2 to 9] | 16 [11 to 21] | 4 [2 to 8]
  Day 15 (N=161, 209, 210) | 99 [96 to 100] | 100 [97 to 100] | 99 [97 to 100]
  Day 36 (N=157, 206, 207) | 100 [98 to 100] | 99 [96 to 100] | 100 [97 to 100]
  Day 57 (157, 204, 204) | 100 [98 to 100] | 97 [93 to 99] | 100 [97 to 100]
  Day 91 (N=152, 206, 204) | 99 [95 to 100] | 85 [79 to 90] | 98 [95 to 99]
  Day 181 (N= 155, 200, 202) | 88 [82 to 92] | 75 [68 to 81] | 89 [84 to 93]
  Day 366 (154, 199, 204) | 76 [68 to 82] | 68 [61 to 74] | 80 [74 to 85]

8. Secondary Outcome: Kinetics of Rabies Immune Response Measured as the RVNA GMCs
Description: To evaluate the kinetics of antibody response to Rabies vaccine, the immunogenicity was measured as the RVNA GMCs on days 1, 8, 15, 36, 57, 91, 181, and 366.
Time Frame: Day 1, 8, 15, 36, 57, 91, 181, and 366
Population: Analysis was done on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv
Number analyzed (Participants) | 166 | 215 | 218
IU/mL
  Day 1 | 0.052 [0.048 to 0.056] | 0.053 [0.049 to 0.056] | 0.054 [0.05 to 0.057]
  Day 8 (N=161, 210, 213) | 0.071 [0.061 to 0.084] | 0.13 [0.12 to 0.16] | 0.076 [0.066 to 0.088]
  Day 15 (N=161, 209, 210), | 21 [17 to 25] | 26 [22 to 30] | 24 [20 to 28]
  Day 36 (N=157, 206, 207) | 14 [12 to 17] | 5.75 [4.95 to 6.67] | 13 [11 to 15]
  Day 57 (N=157, 204, 204) | 10 [8.72 to 12] | 3.01 [2.59 to 3.51] | 9.66 [8.31 to 11]
  Day 91 (N=152, 206, 204) | 4.79 [3.98 to 5.76] | 1.63 [1.39 to 1.91] | 5.04 [4.29 to 5.91]
  Day 181 (N= 155, 200, 202) | 1.86 [1.15 to 2.3] | 1 [0.83 to 1.21] | 2.04 [1.69 to 2.46]
  Day 366 (N=154, 199, 204) | 0.93 [0.75 to 1.16] | 0.82 [0.67 to 1] | 1.14 [0.94 to 1.38]

9. Secondary Outcome: Kinetics of JE Immune Response Measured as Percentage of Subjects With PRNT50 Titers ≥1:10
Description: To evaluate the kinetics of antibody response to JE vaccine, the immunogenicity was measured as the percentage of subjects with PRNT50 titer ≥1:10 on days 1, 15, 22, 36, 57, 91, 181, and 366 (group that received JE vaccine as an accelerated schedule) and days 1, 36, 57, 181, and 366 (group that received JE vaccine as a conventional schedule).
Time Frame: Days 1, 15, 22, 36, 57, 91, 181 and 366
Population: Analysis was done on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | R/JE - Conv | R/JE - Acc | JE - Conv
Number analyzed (Participants) | 165 | 215 | 55
Percentages of subjects
  Day 1 | 1 [0 to 4] | 6 [3 to 10] | 9 [3 to 20]
  Day 15 (N=0, 209, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 99 [96 to 100] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 22 (N=0, 208, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 100 [97 to 100] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 36 (157, 206, 47) | 99 [97 to 100] | 99 [96 to 100] | 100 [92 to 100]
  Day 57 (N=157, 204, 49) | 100 [98 to 100] | 98 [95 to 99] | 100 [93 to 100]
  Day 91 (N=0, 206, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 98 [95 to 99] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 181 (N=155, 200, 49) | 94 [88 to 97] | 98 [94 to 99] | 92 [80 to 98]
  Day 366 (N=154, 199, 48) | 86 [79 to 91] | 94 [90 to 97] | 88 [75 to 95]

10. Secondary Outcome: Kinetics of JE Immune Response Measured as PRNT50 GMTs
Description: To evaluate the kinetics of antibody response to JE vaccine, the immunogenicity was measured as the PRNT50 GMTs on days 1, 15, 22, 36, 57, 91, 181, and 366 (group that received JE vaccine as an accelerated schedule) and days 1, 36, 57, 181, and 366 (group that received JE vaccine as a conventional schedule).
Time Frame: Day 1, 15, 22, 36, 57, 91, 181, and 366 (accelerated schedule) and day 1, 36, 57, 181, and 366 (conventional schedule)
Population: Analysis was done on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | R/JE - Conv | R/JE - Acc | JE - Conv
Number analyzed (Participants) | 165 | 215 | 55
Titers
  Day 1 | 5.13 [4.84 to 5.43] | 5.63 [5.35 to 5.92] | 5.73 [5.2 to 6.33]
  Day 15 (N=0, 209, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 715 [608 to 842] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 22 (0, 208, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 1255 [1068 to 1475] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 36 (N=157, 206, 47) | 292 [247 to 346] | 690 [595 to 801] | 376 [277 to 510]
  Day 57 (N= 157, 204, 49) | 299 [254 to 352] | 372 [322 to 430] | 337 [252 to 451]
  Day 91 (N=0, 206, 0) | NA [NA to NA] — Analysis was not performed in this group at this timepoint. | 228 [192 to 272] | NA [NA to NA] — Analysis was not performed in this group at this timepoint.
  Day 181 (N=155, 200, 49) | 63 [53 to 75] | 151 [130 to 176] | 64 [47 to 87]
  Day 366 (N=154, 199, 48) | 39 [33 to 47] | 117 [100 to 137] | 39 [28 to 54]

11. Secondary Outcome: Number of Subjects Who Reported Solicited Local Adverse Events After Each Rabies Vaccination
Description: Safety was assessed as the number of subjects who reported solicited local adverse events (AEs) after each rabies vaccination given according to accelerated or conventional schedule as follows: from day 1 through day 7 (vaccination on day 1; all Rabies groups), day 4 through day 10 (vaccination on day 4; in R/JE - Acc group only), day 8 through day 14 (vaccination on day 8; all Rabies groups), or day 29 through day 35 (vaccination on day 29; R/JE - Conv and R - Conv groups).
Time Frame: Day 1 through day 7 after each vaccination (on day 1, 4, 8 and 29)
Population: Analysis was done on the solicited safety set, i.e. the subjects in the exposed population who provided postvaccination solicited safety data.
Measure: Number; unit: Number of subjects
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv
Number analyzed (Participants) | 166 | 217 | 220
Number of subjects
  Erythema (day 1 to 7) | 13 | 31 | 28
  Induration (day 1 to 7) | 3 | 16 | 11
  Pain (day 1 to 7) | 43 | 69 | 72
  Erythema (day 4 to 10) | NA — Subjects in this group received placebo at day 4 | 17 | NA — Subjects in this group received placebo at day 4
  Induration (day 4 to 10) | NA — Subjects in this group received placebo at day 4 | 9 | NA — Subjects in this group received placebo at day 4
  Pain (day 4 to 10) | NA — Subjects in this group received placebo at day 4 | 55 | NA — Subjects in this group received placebo at day 4
  Erythema (day 8 to 14) | 8 | 31 | 29
  Induration (day 8 to 14) | 10 | 15 | 17
  Pain (day 8 to 14) | 57 | 87 | 90
  Erythema (day 29 to 35) | 23 | NA — Subjects in this group received placebo at day 29 | 45
  Induration (day 29 to 35) | 18 | NA — Subjects in this group received placebo at day 29 | 32
  Pain (day 29 to 35) | 52 | NA — Subjects in this group received placebo at day 29 | 87

12. Secondary Outcome: Number of Subjects Who Reported Solicited Local AEs After Each JE Vaccination
Description: Safety was assessed as the number of subjects who reported solicited local AEs after each JE vaccination given according to accelerated or conventional schedule as follow: from day 1 through day 7 (vaccination on day 1; all JE groups), day 8 through day 14 (vaccination on day 8; R/JE - Acc group only), or day 29 through day 35 (vaccination on day 29; R/JE - Con and JE - Conv groups).
Time Frame: Day 1 through day 7 after each vaccination (on day 1, 8 and 29)
Population: Analysis was done on the solicited safety set.
Measure: Number; unit: Number of subjects
Arm/Group | R/JE - Conv | R/JE - Acc | JE - Conv
Number analyzed (Participants) | 166 | 217 | 56
Number of subjects
  Erythema (day 1 to 7) | 20 | 30 | 6
  Induration (day 1 to 7) | 13 | 19 | 5
  Pain (day 1 to 7) | 82 | 102 | 26
  Erythema (day 8 to 14) | NA — Subjects in this group didn't receive JE vaccination on day 8. | 18 | NA — Subjects in this group didn't receive JE vaccination on day 8.
  Induration (day 8 to 14) | NA — Subjects in this group didn't receive JE vaccination on day 8. | 12 | NA — Subjects in this group didn't receive JE vaccination on day 8.
  Pain (day 8 to 14) | NA — Subjects in this group didn't receive JE vaccination on day 8. | 60 | NA — Subjects in this group didn't receive JE vaccination on day 8.
  Erythema (day 29 to 35) | 12 | NA — Subjects in this group didn't receive JE vaccination on day 29. | 5
  Induration (day 29 to 35) | 5 | NA — Subjects in this group didn't receive JE vaccination on day 29. | 4
  Pain (day 29 to 35) | 46 | NA — Subjects in this group didn't receive JE vaccination on day 29. | 12

13. Secondary Outcome: Number of Subjects Who Reported Solicited Local AEs After Each Placebo Injection
Description: Safety was assessed as the number of subjects who reported solicited local AEs after each placebo injection given according to accelerated and conventional schedule as follow: from day 1 through day 7 (injection on day 1; R - Conv and JE - Conv groups), day 4 through day 10 (injection on day 4; in R/JE - Conv, R - Conv and JE - Conv groups), day 8 through day 14 (injection on day 8; in R/JE - Conv, R - Conv and JE - Conv groups), and day 29 through day 35 (injection on day 29; R/JE - Acc, R - Con and JE - Conv groups).
Time Frame: Day 1 through day 7 after each injection (day 1, 4, 8 and 29)
Population: Analysis was done on the solicited safety set.
Measure: Number; unit: Number of Subjects
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv
Number analyzed (Participants) | 163 | 213 | 220 | 56
Number of Subjects
  Erythema (day 1 to 7) | NA — Subjects in this group didn't receive placebo at day 1. | NA — Subjects in this group didn't receive placebo at day 1. | 20 | 3
  Induration (day 1 to 7) | NA — Subjects in this group didn't receive placebo at day 1. | NA — Subjects in this group didn't receive placebo at day 1. | 4 | 5
  Pain (day 1 to 7) | NA — Subjects in this group didn't receive placebo at day 1. | NA — Subjects in this group didn't receive placebo at day 1. | 26 | 7
  Erythema (day 4 to 10) | 8 | NA — Subjects in this group didn't receive placebo at day 4. | 13 | 3
  Induration (day 4 to 10) | 1 | NA — Subjects in this group didn't receive placebo at day 4. | 4 | 2
  Pain (day 4 to 10) | 7 | NA — Subjects in this group didn't receive placebo at day 4. | 15 | 3
  Erythema (day 8 to 14) | 1 | NA — Subjects in this group didn't receive placebo at day 8. | 11 | 4
  Erythema (day 8 to 14 after 2nd Placebo dose) | NA — Subjects in this group received only 1 dose of placebo at day 8. | NA — Subjects in this group didn't receive placebo at day 8. | NA — Subjects in this group received only 1 dose of placebo at day 8. | 3
  Induration (day 8 to 14) | 0 | NA — Subjects in this group didn't receive placebo at day 8. | 5 | 1
  Induration (day 8 to 14 after 2nd Placebo dose) | NA — Subjects in this group received only 1 dose of placebo at day 8. | NA — Subjects in this group didn't receive placebo at day 8. | NA — Subjects in this group received only 1 dose of placebo at day 8. | 1
  Pain (day 8 to 14) | 19 | NA — Subjects in this group didn't receive placebo at day 8. | 20 | 3
  Pain (day 8 to 14 after 2nd Placebo dose) | NA — Subjects in this group received only 1 dose of placebo at day 8. | NA — Subjects in this group didn't receive placebo at day 8. | NA — Subjects in this group received only 1 dose of placebo at day 8. | 5
  Erythema (day 29 to 35) | NA — Subjects in this group didn't receive placebo at day 29. | 15 | 15 | 3
  Erythema (day 29 to 35 after 2nd Placebo dose) | NA — Subjects in this group didn't receive placebo at day 29. | 14 | NA — Subjects in this group received only 1 dose of placebo at day 29. | NA — Subjects in this group received only 1 dose of placebo at day 29.
  Induration (day 29 to 35) | NA — Subjects in this group didn't receive placebo at day 29. | 6 | 4 | 1
  Induration (day 29 to 35 after 2nd Placebo dose) | NA — Subjects in this group didn't receive placebo at day 29. | 4 | NA — Subjects in this group received only 1 dose of placebo at day 29. | NA — Subjects in this group received only 1 dose of placebo at day 29.
  Pain (day 29 to 35) | NA — Subjects in this group didn't receive placebo at day 29. | 15 | 28 | 3
  Pain (day 29 to 35 after 2nd Placebo dose) | NA — Subjects in this group didn't receive placebo at day 29. | 19 | NA — Subjects in this group received only 1 dose of placebo at day 29. | NA — Subjects in this group received only 1 dose of placebo at day 29.

14. Secondary Outcome: Number of Subjects Who Reported Solicited Systemic AEs and Other Indicators of Reactogenicity After Each Vaccination
Description: Safety was assessed as the number of subjects who reported solicited systemic AEs and other indicators of reactogenicity after each vaccination given according to accelerated and conventional schedule.
Time Frame: Day 1 through day 7 after each vaccination (day 1, 4, 8 and 29)
Population: Analysis was done on the solicited safety set.
Measure: Number; unit: Number of Subjects
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv
Number analyzed (Participants) | 166 | 217 | 220 | 56
Number of Subjects
  Fatigue (day 1 to 7) | 39 | 56 | 46 | 16
  Headache (day 1 to 7) | 35 | 46 | 38 | 14
  Myalgia (day 1 to 7) | 27 | 55 | 31 | 7
  Arthralgia (day 1 to 7) | 8 | 13 | 7 | 1
  Loss of Appetite (day1 to day 7) | 10 | 8 | 12 | 6
  Nausea (day1 to day 7) | 8 | 7 | 13 | 4
  Body temperature (≥38 °C, day 1 to day 7) | 1 | 2 | 2 | 0
  Analgesic/Antipyretic used (day 1 to day 7) | 11 | 11 | 8 | 3
  Fatigue (day 4 to 10) | 14 | 30 | 33 | 5
  Headache (day 4 to 10) | 17 | 28 | 29 | 3
  Myalgia (day 4 to 10) | 11 | 19 | 14 | 1
  Arthralgia (day 4 to 10) | 1 | 9 | 9 | 0
  Loss of Appetite (day4 to day 10) | 4 | 8 | 9 | 2
  Nausea (day4 to day 10) | 4 | 5 | 8 | 0
  Body temperature (≥38 °C, day 4 to day 10) | 1 | 1 | 2 | 0
  Analgesic/Antipyretic used (day 4 to 10) | 8 | 10 | 15 | 2
  Fatigue (day 8 to 14) | 24 | 47 | 47 | 6
  Headache (day 8 to 14) | 33 | 43 | 41 | 3
  Myalgia (day 8 to 14) | 22 | 41 | 38 | 1
  Arthralgia (day 8 to 14) | 6 | 9 | 13 | 1
  Loss of Appetite (day8 to day 14) | 10 | 14 | 13 | 2
  Nausea (day8 to day 14) | 5 | 14 | 16 | 2
  Body temperature (≥38 °C, day 8 to 14) | 2 | 1 | 5 | 0
  Analgesic/Antipyretic used (day 8 to 14) | 10 | 17 | 20 | 2
  Fatigue (day 29 to 35) | 21 | 29 | 36 | 3
  Headache (day 29 to 35) | 27 | 22 | 40 | 4
  Myalgia (day 29 to 35) | 23 | 15 | 28 | 2
  Arthralgia (day 29 to 35) | 5 | 6 | 14 | 1
  Body temperature (≥38 °C, day 29 to day 35) | 1 | 2 | 1 | 0
  Analgesic/Antipyretic used (day 29 to day 35) | 9 | 10 | 11 | 3
  Loss if appetite (day 29 to day 25) | 2 | 8 | 9 | 2
  nausea (day29 to day 25) | 7 | 12 | 9 | 2

15. Secondary Outcome: Numbers of Subjects Reporting Unsolicited AEs After Any Vaccination From Day 1 Through Day 57
Description: Safety was assessed as the number of subjects who reported unsolicited AEs after any vaccination given according to accelerated and conventional schedule.
Time Frame: Day 1 through Day 57
Population: Analysis was done on the unsolicited safety set, ie, the subjects in the exposed population who provided postvaccination unsolicited safety data.
Measure: Number; unit: Number of subjects
Groups:
- R/JE - Conv: Subjects received Rabies and JE vaccines, conventional schedule, i.e. Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and JE vaccination on day 1 and 29, and placebo on day 8 in the left arm.
- R/JE - Acc: Subjects received Rabies and JE vaccines, accelerated schedule, i.e. Rabies vaccination on days 1, 4, and 8, and placebo on day 29 in the right arm or leg; and JE vaccination on days 1 and 8, and placebo on day 29 in the left arm.
- R - Conv: Subjects received Rabies vaccine, conventional schedule, i.e. Rabies vaccination on days 1, 8, and 29, and placebo on day 4 in the right arm or leg; and placebo on days 1, 8 and 29 in the left arm.
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv
Number analyzed (Participants) | 166 | 217 | 220 | 56
Number of subjects
  Any AE | 69 | 108 | 110 | 29
  SAEs | 2 | 3 | 2 | 3
  AEs leading to premature withdrawal | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected for 7 days after each vaccination. All unsolicited AEs, serious adverse events (SAEs), AEs leading to study and/or treatment withdrawal were collected through day 57. From day 57 to day 366 vaccine-related SAEs were collected.
Description: Solicited adverse events were collected by systematic assessment, unsolicited AEs by non-systematic assessment. SAEs analysis was done one the unsolicited safety set, other AEs analysis was done on the overall safety set.
Arm/Group | R/JE - Conv | R/JE - Acc | R - Conv | JE - Conv
Serious Adverse Events (participants affected / at risk) | 2/166 | 3/217 | 2/220 | 3/56
Other Adverse Events (participants affected / at risk) | 138/166 | 186/217 | 185/220 | 45/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R/JE - Conv (N=166) | R/JE - Acc (N=217) | R - Conv (N=220) | JE - Conv (N=56)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
EYELID OEDEMA (Eye disorders) | 0 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OVARIAN GERM CELL TERATOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R/JE - Conv (N=166) | R/JE - Acc (N=217) | R - Conv (N=220) | JE - Conv (N=56)
NAUSEA (Gastrointestinal disorders) | 19 | 31 | 35 | 9
FATIGUE (General disorders) | 54 | 93 | 84 | 19
INJECTION SITE ERYTHEMA (General disorders) | 48 | 73 | 85 | 13
INJECTION SITE INDURATION (General disorders) | 29 | 43 | 48 | 10
INJECTION SITE PAIN (General disorders) | 115 | 146 | 131 | 31
NASOPHARYNGITIS (Infections and infestations) | 22 | 33 | 32 | 7
DECREASED APPETITE (Metabolism and nutrition disorders) | 19 | 24 | 27 | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 29 | 31 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 50 | 75 | 60 | 10
HEADACHE (Nervous system disorders) | 63 | 94 | 95 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less